CLINICAL TRIAL: NCT03453840
Title: Extended Duration Artemether-lumefantrine Treatment for Malaria in Children
Acronym: EXALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Yale University (Other); Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22578; 2R01HD068174-06A1 (NIH)
Record Dates: First submitted 2017-12-22; First posted 2018-03-05 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: malaria; HIV; Children; Efavirenz; artemether; lumefantrine
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: This is a prospective multi-site study accomplished through a randomized design where children will be randomized to either 3-day or 5-day AL regimen and then for subsequent episodes of malaria, should they occur..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HIV-infected 3-day AL (Active Comparator): Standard 3-day twice daily (BID) regimen of artemether-lumefantrine for uncomplicated malaria, given over 4 days (Study Days 0, 1, 2 and 3) so that sampling will begin in the morning of day 3. These participants are HIV-infected and stabilized on EFV-based ART.
  Interventions: Drug: Artemether-lumefantrine
- HIV-infected 5-day AL (Experimental): Extended 5-day BID regimen of artemether-lumefantrine, given over 6 days (Study Days 0, 1, 2, 3, 4, and 5) so that sampling will begin in the morning of day 5. These participants are HIV-infected and stabilized on EFV-based ART.
  Interventions: Drug: Artemether-lumefantrine
- HIV-uninfected 3-day AL (Active Comparator): Standard 3-day BID regimen of artemether-lumefantrine for uncomplicated malaria, given over 4 days (Study Days 0, 1, 2 and 3) so that sampling will begin in the morning of day 3. These participants are HIV-uninfected.
  Interventions: Drug: Artemether-lumefantrine
- HIV-uninfected 5-day AL (Experimental): Extended 5-day BID regimen of artemether-lumefantrine, given over 6 days (Study Days 0, 1, 2, 3, 4, and 5) so that sampling will begin in the morning of day 5. These participants are HIV-uninfected.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Children will receive the dispersible formulation of AL which contains 20 mg artemether, 120 mg of lumefantrine (Coartem® Dispersible). Weight-based dosing will be as below: <15kg, 1tablet; 15-25kg, 2 tablets; 25-35kg, 3 tablets; >=35kg, 4 tablets.
  Other Names: Coartem, AL

SUMMARY:
This project determines the pharmacokinetic/pharmacodynamic (PK/PD) of an extended artemether-lumefantrine (AL) dosing regimen in HIV-infected children on efavirenz (EFV)-based antiretroviral therapy (ART) that is designed to improve the PK exposure and treatment efficacy of this artemisinins-based combination therapy (ACT) regimen. Our overarching goal is to inform the best treatment guidelines for young children in Africa. HIV-infected and HIV-uninfected children were enrolled for intensive PK studies, as well as additional children for population PK studies to enhance association analyses with clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective multi-site study to evaluate the PK/PD of extended duration AL in HIV-infected children on EFV-based ART and HIV-uninfected children not on ART. AL is the first-line treatment for malaria in Uganda. No change in standard of care treatment was made for the purposes of this study except for the extension of AL to 5-day dosing. This study enrolled a) HIV-infected children, and b) HIV-uninfected children. All participants may be enrolled through Tororo District Hospital (TDH) or Masafu General Hospital (MGH) in Busia, or other referral centers the area. we used a design where children were randomized to either 3-day or 5-day AL and then for subsequent episodes of malaria, should they occur. Conservatively, assuming each enrolled child participates for only a single episode of malaria, up to 60 (30 HIV-infected on 3-day and 30 HIV-infected on 5-day) and 100 (50 HIV-uninfected on 3-day and 50 HIV-uninfected on 5-day) subjects were enrolled for each of the intensive study groups. 16 (9 HIV-infected on 3-day and 7 HIV-infected on 5-day) and 120 (60 HIV-uninfected on 3-day and 60 HIV-uninfected on 5-day) subjects were enrolled for each of the population study groups. Enrollment of HIV-infected subjects for population PK study groups was not halted due to the lack of HIV-infected children in the study area. Comparisons of AL PK exposure were made among and between a) HIV-infected children with malaria receiving EFV-based ART and b) HIV-uninfected children who are not on ART. Comparisons were based on an intensive PK design for AL area under the concentration-time curve (AUC) estimations.

ELIGIBILITY:
Inclusion Criteria:

1, All participants:

1. Residency within 60 km of the study clinics either at TDH or at MGH
2. Agreement to come to clinic for all follow-up clinical and PK evaluations
3. Provision of informed consent
4. Weight ≥6 kg
5. Presentation with uncomplicated falciparum malaria as indicated by positive smear for malaria parasites along with clinical evidence of infection (fever or history of fever in the past 24 hours)
6. Willingness to undergo intensive PK sampling and/or population PK sampling during episode(s) of malaria.

2 HIV-infected participants:

1. Confirmed HIV infection (positive rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
2. On stable EFV-based ART for at least 10 days prior to enrollment
3. Age 3 years to 18 years

3 HIV-uninfected participants:

1. Confirmed HIV negative test (negative rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
2. Age 6 months to 18 years

Exclusion Criteria:

1. History of significant comorbidities such as malignancy, active tuberculosis or other World Health Organization (WHO) stage 4 disease
2. Current infection with non-P. falciparum species
3. Receipt of any medications known to affect CYP450 metabolism (except ART) within 14 days of study enrollment (see 4.2.2)
4. Hemoglobin < 7.0 g/dL
5. For the population PK study, prior treatment for malaria within 14 days of enrollment
6. For the intensive PK study, prior treatment for malaria within 28 days of enrollment
7. Signs or evidence of complicated malaria, defined as unarousable coma or any two of the following symptoms: Recent febrile convulsions, altered consciousness, lethargy, unable to drink, unable to stand/sit due to weakness, severe anemia (Hb < 5.0 gm/dL), respiratory distress, jaundice (see Appendix D)
8. History of toxicity to AL

The following medications are disallowed within 3 weeks prior to receiving study drug:

* Carbamazepine
* Clarithromycin
* Erythromycin (oral)
* Ketoconazole
* Phenobarbital
* Phenytoin
* Rifabutin
* Rifampin
* Halofantrine
* Any other medication known to significantly affect CYP450 metabolism.
* Grapefruit juice should be avoided during the study due to its potential effects on CYP3A4.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Pharm. D, Principal Investigator — University of California, San Francisco; Sunil Parikh, M.D., MPH, Principal Investigator — Yale University School of Public Health
Locations (2):
- Uganda (2):
  - MGH campus, Busia
  - IDRC- Tororo Research Clinic and Tororo District Hospital, Tororo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Whalen ME, Kajubi R, Goodwin J, Orukan F, Colt M, Huang L, Richards K, Wang K, Li F, Mwebaza N, Aweeka FT, Parikh S. The Impact of Extended Treatment With Artemether-lumefantrine on Antimalarial Exposure and Reinfection Risks in Ugandan Children With Uncomplicated Malaria: A Randomized Controlled Trial. Clin Infect Dis. 2023 Feb 8;76(3):443-452. doi: 10.1093/cid/ciac783. PMID 36130191
- [Result] Whalen ME, Kajubi R, Goodwin J, Orukan F, Colt M, Huang L, Richards K, Hoffmann TJ, Aweeka FT, Parikh S, Mwebaza N. Extended Treatment Duration of Artemether-Lumefantrine in Ugandan Children with HIV on Efavirenz-Based Antiretroviral Therapy: A Randomized Controlled Pharmacokinetic and Pharmacodynamic Trial. J Clin Pharmacol. 2025 Jul;65(7):909-922. doi: 10.1002/jcph.6193. Epub 2025 Jan 24. PMID 39853752
- [Derived] Goodwin J, Kajubi R, Wang K, Li F, Wade M, Orukan F, Huang L, Whalen M, Aweeka FT, Mwebaza N, Parikh S. Persistent and multiclonal malaria parasite dynamics despite extended artemether-lumefantrine treatment in children. Nat Commun. 2024 May 7;15(1):3817. doi: 10.1038/s41467-024-48210-7. PMID 38714692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on 2/21/2018 and ended on 07/23/2019 and last follow up date was 09/03/2019. Study location was at Masafu General Hospital. Intensive PK recruitments were completed for all 4 arms: HIV negative 3-day and 5-day arm (n=50 each), HIV positive 3-day and 5-day arm (n=30). Population PK recruitments reached the target for HIV negative arms (n=60 each), but not for HIV-positive arms, because of the lack of HIV positive patients in the study sites.
Period: Overall Study
Arm/Group | HIV-infected 3-day AL | HIV-infected 5-day AL | HIV-uninfected 3-day AL | HIV-uninfected 5-day AL
Started | 39 (The 1st PID (50017) was recruited on 3/26/2018 but withdrawn due to mixed infection. 1st completed PID50039 was recruited on 5/21/2018.) | 37 (The 1st intensive PID50019 enrolled on 4/4/2018.) | 115 | 114 (1st participant enrolled on 2/21/2018 did not complete the study and the 1st completed one was enrolled on 3/01/2018)
Completed | 35 (n=30 (intensive) and 5(pop). The last intensive PID 50307 enrolled on 11/27/2019 completed on 1/08/2020. POP PK completed on 1/9/2020 (PID50309).) | 36 (n=30(intensive) and 6(pop). The last intensive PID50304 enrolled on 11/20/2019 completed on 1/02/2020. POP PK completed on 9/3/2019 (PID50283).) | 110 (last intensive PK PID (50114) enrolled on 9/19/2018 and completed follow up on 10/31/2018. Pop PK completed on 8/29/2019 (PID50281).) | 110 (The last intensive PK participant (50123) was not completed follow up due to treatment failure and ended on 11/5/2018. The last follow up date for intensive PK was 11/09/2018 (PID50120). Pop PK completed on 8/28/2019 (PID50278))
Not Completed | 4 | 1 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Eligible HIV negative participant age range is 6 months to 18 years and HIV positive participant age range 3-18 years.
Groups:
- HIV-infected 3-day AL Intensive PK: Standard 3-day twice daily (BID) regimen of artemether-lumefantrine for uncomplicated malaria, given over 4 days (Study Days 0, 1, 2 and 3) so that sampling will begin in the morning of day 3. These participants are HIV-infected and stabilized on EFV-based ART.
  Artemether-lumefantrine: Children will receive the dispersible formulation of AL which contains 20 mg artemether, 120 mg of lumefantrine (Coartem® Dispersible). Weight-based dosing will be as below: <15kg, 1tablet; 15-25kg, 2 tablets; 25-35kg, 3 tablets; >=35kg, 4 tablets.
- HIV-infected 5-day AL Intensive PK: Extended 5-day BID regimen of artemether-lumefantrine, given over 6 days (Study Days 0, 1, 2, 3, 4, and 5) so that sampling will begin in the morning of day 5. These participants are HIV-infected and stabilized on EFV-based ART.
  Artemether-lumefantrine: Children will receive the dispersible formulation of AL which contains 20 mg artemether, 120 mg of lumefantrine (Coartem® Dispersible). Weight-based dosing will be as below: <15kg, 1tablet; 15-25kg, 2 tablets; 25-35kg, 3 tablets; >=35kg, 4 tablets.
- Total: Total of all reporting groups
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL | HIV-uninfected 5-day AL | Total
Number analyzed (Participants) | 35 | 36 | 114 | 113 | 298
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.5 [7.71 to 14.25] | 10.4 [7.13 to 13.4] | 5.3 [4.1 to 7.9] | 5.9 [4.1 to 8.0] | 6.2 [4.3 to 9.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 64 | 60 | 160
  Male | 14 | 21 | 50 | 53 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 35 | 36 | 114 | 113 | 298
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 35 | 36 | 114 | 113 | 298
Weight [Median (Inter-Quartile Range); unit: kg] | 28.4 [22.0 to 35.5] | 25.8 [21.2 to 30.1] | 17.3 [15.1 to 23.0] | 19.1 [15.4 to 22.6] | 20.2 [15.8 to 26.5]

OUTCOME MEASURES:

1. Primary Outcome: AUC0-21d
Description: Area under the plasma concentration versus time curve (AUC) from time 0 to day 21 for lumefantrine
Time Frame: Study day 0-day21
Population: Intensive PK participants only. Population PK participants are excluded here.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ug/mL
Groups:
- HIV-uninfected 3-day AL Intensive PK: Standard 3-day BID regimen of artemether-lumefantrine for uncomplicated malaria, given over 4 days (Study Days 0, 1, 2 and 3) so that sampling will begin in the morning of day 3. These participants are HIV-uninfected.
  Artemether-lumefantrine: Children will receive the dispersible formulation of AL which contains 20 mg artemether, 120 mg of lumefantrine (Coartem® Dispersible). Weight-based dosing will be as below: <15kg, 1tablet; 15-25kg, 2 tablets; 25-35kg, 3 tablets; >=35kg, 4 tablets.
- HIV-uninfected 5-day AL Intensive PK: Extended 5-day BID regimen of artemether-lumefantrine, given over 6 days (Study Days 0, 1, 2, 3, 4, and 5) so that sampling will begin in the morning of day 5. These participants are HIV-uninfected.
  Artemether-lumefantrine: Children will receive the dispersible formulation of AL which contains 20 mg artemether, 120 mg of lumefantrine (Coartem® Dispersible). Weight-based dosing will be as below: <15kg, 1tablet; 15-25kg, 2 tablets; 25-35kg, 3 tablets; >=35kg, 4 tablets.
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
hr*ug/mL | 144 [114 to 182] | 205 [151 to 279] | 259 [222 to 302] | 318 [274 to 370]

2. Primary Outcome: Recurrent Parasitemia Following Treatment by Day 42 (Recrudescence or New Infection)
Description: Recurrent malaria determined by microscopy (thick blood smears), loop mediated isothermal amplification (LAMP), or rapid diagnostic test (RDT).
Time Frame: up to study day 42
Population: All participants including intensive and population PK participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected 3-day AL | HIV-infected 5-day AL | HIV-uninfected 3-day AL | HIV-uninfected 5-day AL
Number analyzed (Participants) | 36 | 36 | 114 | 113
Participants | 19 | 18 | 80 | 66

3. Primary Outcome: AUC0-8h for Artemether
Description: Area under the plasma concentration versus time curve (AUC) from 0 to 8hr post last dose for artemether (ARM)
Time Frame: 0-8hr
Population: Intensive PK participants only, so the participant number here is different from the numbers in the participant flow module, which includes both intensive and population PK participants.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
hr*ng/mL | 64.0 [45.5 to 90] | 71.7 [54.8 to 93.8] | 95.8 [77.5 to 118] | 78.6 [61.3 to 101]

4. Primary Outcome: AUC0-8h for Dihydroartemisinin
Description: Area under the plasma concentration versus time curve (AUC) from time 0 to 8hr post last dose for Dihydroartemisinin (DHA)
Time Frame: 0-8hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: hr.ng/mL
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
hr.ng/mL | 109 [83.9 to 142] | 95.8 [69.7 to 132] | 241 [216 to 269] | 229 [202 to 261]

5. Primary Outcome: Cmax for Lumefantrine
Description: Maximal concentration post last dose for lumefantrine
Time Frame: 0-21 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
ng/mL | 5065 [3894 to 6589] | 6027 [4253 to 8543] | 7236 [6023 to 8692] | 8450 [7085 to 10079]

6. Primary Outcome: Cmax for Artemether
Description: Maximal concentration post last dose for artemether
Time Frame: 0-8hr
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
ng/mL | 22.4 [15.3 to 32.8] | 23.0 [16.4 to 32.3] | 32.5 [25.4 to 41.5] | 27.3 [20.5 to 36.3]

7. Primary Outcome: Cmax for Dihydroartemisinin
Description: Maximal concentration post last dose for dihydroartimisinin (DHA)
Time Frame: 0-8hr
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HIV-infected 3-day AL Intensive PK | HIV-infected 5-day AL Intensive PK | HIV-uninfected 3-day AL Intensive PK | HIV-uninfected 5-day AL Intensive PK
Number analyzed (Participants) | 30 | 30 | 50 | 50
ng/mL | 43.8 [33.5 to 57.2] | 34.9 [24.6 to 49.4] | 89.0 [77.4 to 102] | 87.9 [75.8 to 102]

8. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: We recorded participants tolerance of AL using the NIH Division of AIDS Adult and Pediatric Toxicity Tables.
Time Frame: study day 0-42
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected 3-day AL | HIV-infected 5-day AL | HIV-uninfected 3-day AL | HIV-uninfected 5-day AL
Number analyzed (Participants) | 35 | 36 | 114 | 113
Participants | 0 | 0 | 2 | 0

9. Other Pre Specified Outcome: Relationship Between Drug Resistance and Treatment Failure
Description: drug resistance will be accessed by molecular markers. Polymorphic markers will be typed using capillary electrophoresis.
Time Frame: study day 0-42
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Metabolomic Measurements in HIV Infected vs HIV Uninfected Children
Description: Small-molecule metabolites, including metabolic intermediates, hormones and other signaling molecules, and secondary metabolites will be measured in plasma and reported as fold-change (e.g. infected vs uninfected). This is an exploratory study. The multiple measurements could be aggregated to fold-change.
Time Frame: study day 0-42
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Height-for-age (HFA) Associations With PK
Description: chronic protein-calorie malnutrition resulting in slow linear growth (decreased height-for-age: HFA; stunting).
Time Frame: study day 0
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Diagnostic Sensitivity of LAMP, HS-RDT, and Microscopy for the Detection of Recurrent Parasitemia
Description: Using Loop-mediated isothermal amplification (LAMP), highly sensitive Rapid Diagnostic Test (HS-RDT), and microscope to diagnose recurrent parasitemia.
  study day 0-42
Time Frame: study day 0-42
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Weight-for-height (WFH) Associations With PK
Description: acute protein-calorie malnutrition resulting in weight loss or slow weight gain (decreased weight-for-height: WFH; wasting).
Time Frame: study day 0
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Weight-for-age (WFA) Associations With PK
Description: weight-for-age is an indicator of nutrition status and decreased weight-for-age reflects the combination of chronic and acute protein-calorie malnutrition.
Time Frame: study day 0
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Prevalence of Gametocytemia
Description: At varied time points, blood smears for the determination of parasitemia will be obtained following treatment in 3-day vs 5-day AL regimens.
Time Frame: study day 0-42
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: days 0 to 42
Arm/Group | HIV-infected 3-day AL | HIV-infected 5-day AL | HIV-uninfected 3-day AL | HIV-uninfected 5-day AL
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/114 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 2/114 | 0/113
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/114 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-infected 3-day AL (N=35) | HIV-infected 5-day AL (N=36) | HIV-uninfected 3-day AL (N=114) | HIV-uninfected 5-day AL (N=113)
hypoglycemia (Blood and lymphatic system disorders) | NA | NA | 1 (1) | NA — hypoglycemia on day 26
anemia (Blood and lymphatic system disorders) | NA | NA | 1 (1) | NA — grade 4 anemia on day 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03453840/Prot_SAP_002.pdf
  • Informed Consent Form: Informed Consent Forms (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03453840/ICF_003.pdf
  • Informed Consent Form: Assent and consent for future use of specimen (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03453840/ICF_004.pdf